CLINICAL TRIAL: NCT01386528
Title: An Open-label, Multi-centre, Un-controlled Trial to Assess Efficacy and Safety of NNC-0156-0000-0009 During Surgical Procedures in Patients With Haemophilia B
Brief Title: Efficacy and Safety of NNC-0156-0000-0009 During Surgical Procedures in Subjects With Haemophilia B
Acronym: paradigm™ 3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN7999-3773; 2010-023070-40 (EudraCT Number); U1111-1121-4554 (Other: WHO)
Record Dates: First submitted 2011-06-30; First posted 2011-07-01 (Estimated); Results first posted 2017-07-24 (Actual); Last update posted 2017-08-23 (Actual); Status verified 2017-07

CONDITIONS: Congenital Bleeding Disorder; Haemophilia B
MeSH Terms: conditions — Hemophilia B | interventions — nonacog beta pegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients enrolled in trial (Experimental): New patients will be included as well as transferred patients from Paradigm™ 2 or Paradigm™ 4 trial
  Interventions: Drug: nonacog beta pegol

INTERVENTIONS:
Drug: nonacog beta pegol — The patients will receive nonacog beta pegol at screening just prior to and during surgical intervention, administered intravenously (into the vein).
  Other Names: NNC-0156-0000-0009

SUMMARY:
This trial is conducted in Africa, Asia, Europe and the United States of America (USA).

The aim of the trial is to evaluate the safety and efficacy of NNC-0156-0000-0009 (nonacog beta pegol) during surgical procedures in patients with haemophilia B.

ELIGIBILITY:
Inclusion Criteria:

* Patients with haemophilia B with a FIX activity below or equal to 2%
* Male patients with moderately severe or severe congenital haemophilia B with a FIX activity below or equal to 2% according to medical records
* History of at least 150 exposure days to other FIX products
* Scheduled major surgery

Exclusion Criteria:

* Known history of FIX (coagulation factor nine) inhibitors based on existing medical records, laboratory report reviews and patient and LAR (legal acceptable representative) interviews
* Current FIX (coagulation factor nine) inhibitors above or equal to 0.6 Bethesda Units (central laboratory)
* Previous arterial thrombotic events (e.g. myocardial infarction and intracranial thrombosis) or previous deep venous thrombosis or pulmonary embolism (as defined by available medical records)
* ALT (alanine aminotransferase) 3 times the upper limit of normal reference ranges at screening (central laboratory)
* Immune modulating or chemotherapeutic medication

Ages: 13 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-06-07 (Actual); Primary Completion 2013-12-01 (Actual); Study Completion 2013-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (40):
- United States (7):
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, San Francisco, California
  - Novo Nordisk Investigational Site, Washington D.C., District of Columbia
  - Novo Nordisk Investigational Site, Augusta, Georgia
  - Novo Nordisk Investigational Site, Iowa City, Iowa
  - Novo Nordisk Investigational Site, Syracuse, New York
  - Novo Nordisk Investigational Site, Houston, Texas
- Novo Nordisk Investigational Site, Vienna, Austria
- France (2):
  - Novo Nordisk Investigational Site, Le Kremlin-Bicêtre
  - Novo Nordisk Investigational Site, Lyon
- Germany (4):
  - Novo Nordisk Investigational Site, Bonn
  - Novo Nordisk Investigational Site, Duisburg
  - Novo Nordisk Investigational Site, Giessen
  - Novo Nordisk Investigational Site, Hanover
- Novo Nordisk Investigational Site, Athens, Greece
- Italy (2):
  - Novo Nordisk Investigational Site, Florence
  - Novo Nordisk Investigational Site, Milan
- Japan (6):
  - Novo Nordisk Investigational Site, Kashihara-shi, Nara
  - Novo Nordisk Investigational Site, Kawasaki-shi, Kanagawa
  - Novo Nordisk Investigational Site, Nagoya-shi, Aichi
  - Novo Nordisk Investigational Site, Nishinomiya-shi
  - Novo Nordisk Investigational Site, Suginami-ku, Tokyo
  - Novo Nordisk Investigational Site, Tokyo
- Novo Nordisk Investigational Site, Kuala Lumpur, Malaysia
- Novo Nordisk Investigational Site, Utrecht, Netherlands
- Novo Nordisk Investigational Site, Skopje, North Macedonia
- Novo Nordisk Investigational Site, Timișoara, Timiș County, Romania
- Novo Nordisk Investigational Site, Parktown Johannesburg, Gauteng, South Africa
- Spain (2):
  - Novo Nordisk Investigational Site, Madrid
  - Novo Nordisk Investigational Site, Valencia
- Novo Nordisk Investigational Site, Taipei, Taiwan
- Novo Nordisk Investigational Site, Bangkok, Thailand
- Turkey (Türkiye) (3):
  - Novo Nordisk Investigational Site, Ankara
  - Novo Nordisk Investigational Site, Kayseri
  - Novo Nordisk Investigational Site, Konya
- United Kingdom (5):
  - Novo Nordisk Investigational Site, Basingstoke
  - Novo Nordisk Investigational Site, Cardiff
  - Novo Nordisk Investigational Site, London
  - Novo Nordisk Investigational Site, Manchester
  - Novo Nordisk Investigational Site, Oxford

REFERENCES:
- [Background] Escobar M, Colberg T, Karim F, Caliskan U, Chowdary P, Giangrande P, Giermasz A, Mancuso ME, Serban M, Tsay W, Zak M and Mahlangu J. Perioperative hemostatic management of major surgery in hemophilia B with long-acting recombinant glycopegylated factor IX: results from the paradigm™3 clinical trial. Journal of Thrombosis and Haemostasis (Abstracts) 2015; 13 (Supplement S2): 1-997 [OR348]
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 10 sites in 8 countries : Italy (1 site), Malaysia (1 site), Romania (1 site), South Africa (1 site), Taiwan (1 site), Turkey (1 SIte), UK (2 sites), US (2 sites).
Pre-assignment Details: Patients enrolled in the present trial were recruited from the pivotal trial (NN7999-3747) or the extension trial (NN7999-3775). In addition, new patients were recruited into the present trial.
Groups:
- Nonacog Beta Pegol: New patients as well as transferred patients from the pivotal trial (NN7999-3747) or the extension trial(NN7999-3775) received nonacog beta pegol at screening and followed a preventive treatment regimen with nonacog beta pegol until one week before the day of surgery. No more than 4 hours prior to the planned surgical procedure, all patients received a single bolus injection of 80 U/kg of nonacog beta pegol. Postoperatively, the patients received fixed doses of 40 U/kg repeated at the investigator's discretion aiming for no less than the FIX levels recommended by the World Federation of Hemophilia. Nonacog beta pegol was administered intravenously. The new patients were dosed once with 40 U/kg nonacog beta pegol at screening.From the day after surgery (Day 1) and through Day 6, nonacog beta pegol dosing was adjusted to aim for a FIX activity level of approximately 0.50 U/mL.
Period: Overall Study
Arm/Group | Nonacog Beta Pegol
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set consists of all patients exposed to nonacog beta pegol.
Arm/Group | Nonacog Beta Pegol
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 39 (12.6) [15 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Haemostatic Effect During Surgery Evaluated by the Four-point Response Scale (Excellent, Good, Moderate, Poor)
Description: Haemostatic effect during surgery was evaluated immediately after surgery (last stitch) using a fourpoint response scale:
  - Four-point response scale: Excellent, good, moderate, poor. The evaluation was done by the surgeon, anaesthesiologist and/or investigator based on experience as follows:
  1. Excellent: Better than expected/predicted in this type of procedure.
  2. Good: As expected in this type of procedure.
  3. Moderate: Less than optimal for the type of procedure but haemostatic response maintained without change of treatment regimen.
  4. Poor: Bleeding due to inadequate therapeutic response with adequate dosing, change of regimen required.
Time Frame: At the day of surgery
Population: The full analysis set consisted of all patients exposed to nanacog beta pegol.
Measure: Number; unit: Haemostatic responses
Arm/Group | Nonacog Beta Pegol
Number analyzed (Participants) | 13
Haemostatic responses
  Excellent | 10
  Good | 3
  Moderate | 0
  Poor | 0

2. Secondary Outcome: Consumption of NNC-0156-0000-0009 (U/kg Body Weight)
Description: Mean consumption of nonacog beta pegol (U/kg) used for treatment per patient before surgery, during surgery (the time from knife to skin until last stitch) and post-operative period.
Time Frame: During surgery (the time from knife to skin until last stitch) and post-operative period (day 1 to day 13)
Population: The full analysis set consisted of all patients exposed to nanacog beta pegol.
Measure: Mean (Standard Deviation); unit: U/Kg
Arm/Group | Nonacog Beta Pegol
Number analyzed (Participants) | 13
U/Kg | 328.2 (113.1)

3. Secondary Outcome: Transfusion Requirements (Fulfilling Transfusion Criteria)
Description: Mean quantity of transfusion during surgery (the time from knife to skin until last stitch) and the postoperative period (Day 1-13).None of the patients required transfusions beyond Day 6 hence no values presented for days 7-13.
Time Frame: during surgery (the time from knife to skin until last stitch) and post-operative period (day 1 to day 13)
Population: The full analysis set consisted of all patients exposed to nanacog beta pegol.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Nonacog Beta Pegol
Number analyzed (Participants) | 13
mL
  During surgery | 275 (35.4)
  Post surgery through day 6 | 266.7 (28.9)

4. Secondary Outcome: Haemoglobin Pre- and Post-surgery Start
Description: The mean pre-surgery and post surgery haemoglobin level.
Time Frame: 0, 1 hour, 24 hours.
Population: The full analysis set consisted of all patients exposed to nanacog beta pegol.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Nonacog Beta Pegol
Number analyzed (Participants) | 13
mmol/L
  prior to surgery | 8.98 (0.67)
  1 hour post-surgery | 8.37 (0.78)
  24 hours post surgery | 7.99 (1.13)

5. Secondary Outcome: Incidence of Adverse Events (AEs)
Description: The number of adverse events per patient years of exposure, reported during the trial period. Number is the only available option here, the data presented are rate of AEs.
Time Frame: during the trial period (2-8 weeks prior to day of surgery (transferred subjects) or 2-4 weeks prior to day of surgery (new subjects) until 4 weeks after post-operative period (day 1 to day 13)
Population: The safety analysis set consisted of all patients exposed to nanacog beta pegol.
Measure: Number; unit: events per patient year of exposure
Arm/Group | Nonacog Beta Pegol
Number analyzed (Participants) | 13
events per patient year of exposure | 12.12

6. Secondary Outcome: Incidence of Serious Adverse Events (SAE)
Description: The number of serious adverse events per patient years of exposure, reported during the trial period. Number is the only available option here, the data presented are rate of AEs.
Time Frame: as for outcome 5
Population: The safety analysis set consisted of all patients exposed to nanacog beta pegol.
Measure: Number; unit: Events per patient year of exposure
Arm/Group | Nonacog Beta Pegol
Number analyzed (Participants) | 13
Events per patient year of exposure | 0

7. Secondary Outcome: Incidence of Inhibitors Against FIX (Coagulation Factor Nine)
Description: Number of patients with inhibitory antibodies
Time Frame: During the trial period (2-8 weeks prior to day of surgery (transferred subjects) or 2-4 weeks prior to day of surgery (new subjects) and every 4 weeks after post-operative period (day 1 to day 13)
Population: The full analysis set consisted of all patients exposed to nanacog beta pegol.
Measure: Number; unit: patients
Arm/Group | Nonacog Beta Pegol
Number analyzed (Participants) | 13
patients | 0

ADVERSE EVENTS:
Time Frame: AEs from screening visit (day 0) and until post treatment follow-up period. Patients not continuing in the extension trial attended a follow-up visit 4 weeks ± 2 weeks after the last dose of nonacog beta pegol.
Description: The safety analysis set consisted of all patients exposed to nanacog beta pegol.
Arm/Group | Nonacog Beta Pegol
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 9/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nonacog Beta Pegol (N=13)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 1 (1)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 1 (1)
Face oedema (General disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Oral mucosal erythema (Gastrointestinal disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Serum ferritin increased (Investigations) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This is a single armed study having no comparator.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
"At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property"